CLINICAL TRIAL: NCT06011538
Title: The WISH Trial (Web-based Versus Standard Information for Same Day Hysterectomy)
Brief Title: Web-based Versus Standard Information for Same Day Hysterectomy (WISH)
Acronym: WISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BirminghamWCNHSFT
Record Dates: First submitted 2023-08-09; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hysterectomy; LAP
Keywords: Same day discharge; Laparoscopic hysterectomy; Educational platform; Enhanced recovery

STUDY DESIGN:
Intervention Model Description: To evaluate the potential efficacy of additional on-line, patient education for SDD LH in achieving SDD compared to standard information giving. In addition, the utility and acceptability of patient information will be assessed as well as the impact on patient satisfaction and recovery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-line SDD LH website resource (intervention) (Experimental): Patients allocated the experimental arm will be provided with the link to the SDD LH patient information website (https://www.mydaycasehysterectomy.com).The option of this educational material will be in addition to the standard verbal and written patient information provided by the BWCH.
  Interventions: Other: On-line, multi-media information on a specifically designed website for Same Day Discharge following Laparoscopic Hysterectomy
- Standard practice for information provision (control) (Active Comparator): Patients allocated the control group will receive standard BWCH information only.
  Interventions: Other: On-line, multi-media information on a specifically designed website for Same Day Discharge following Laparoscopic Hysterectomy

INTERVENTIONS:
Other: On-line, multi-media information on a specifically designed website for Same Day Discharge following Laparoscopic Hysterectomy — A patient educational website that provides clear, easily accessible, patient friendly information explaining what SDD after laparoscopic hysterectomy is, why SDD may be beneficial and what to expect from decision for surgery, through to the admission to hospital and immediate, short and long term recovery.

SUMMARY:
Objectives: To evaluate the potential utility and efficacy of additional on-line, patient education resource for same day discharge following laparoscopic hysterectomy (SDD LH) compared to standard information resources alone

Trial Design: A pilot, parallel, open, single centre, randomised controlled trial

Participant Population and Sample Size: 40 women undergoing SDD LH for a benign reason

Eligibility Criteria: Women with gynaecological conditions requiring a laparoscopic hysterectomy (LH) and who are suitable for same day discharge (SDD).

Interventions: An online patient education website resource and the comparator is standard practice for provision of patient information (written and verbal).

Outcome Measures:

Primary

* Compliance with SDD Secondary
* In Hospital:

  o Surgical details / complexity / intraoperative and post-operative serious adverse events (SAEs) according to the Clavien-Dindo system grade II-IV which is a widely used index for the classification of surgical complications [case notes and electronic patient record], and time to discharge
* 6 weeks:

  * Satisfaction, acceptability and utility of patient education / information provided (bespoke patient questionnaire; Likert scales)
  * Satisfaction with care after LH (6-point Likert)
  * Generic quality of life at 6 weeks post-surgery (EuroQol-5D-5L and VAS);
  * Contact with Community & Clinical Care Services i.e. outpatients or emergency visits, re-presentations / re-admissions to hospital (Case report form [CRF], case notes, electronic patient record)
  * Serious Adverse Events (CRF, case notes, electronic patient record)
  * Time from surgery to resumption of usual activities using the PROMIS-SF (Patient-Reported Outcomes Measurement Information System Physical Function) questionnaire (Modified items / response categories)
* 12 weeks:

  * Time from surgery to resumption of usual activities using the PROMIS-SF (Patient-Reported Outcomes Measurement Information System Physical Function) questionnaire (Modified items / response categories) Time to return to work (if working)

DETAILED DESCRIPTION:
Aim:

To evaluate the potential efficacy of additional on-line, patient education for SDD LH in achieving SDD compared to standard information giving. In addition, the utility and acceptability of patient information will be assessed as well as the impact on patient satisfaction and recovery.

Objectives:

The investigators aim to assess various aspects of trial management and design. In order to achieve this, the objectives of the pilot randomised controlled trial (RCT) will be split into:

* Process Objectives

  * To determine the proportion of eligible women that are screened and meet the inclusion criteria
  * To determine the proportion of eligible women that agree to be randomised
  * To determine the robustness of proposed data collection tools; completion and return rates
* Clinical Objectives

  * To determine the appropriateness of the outcome measures
  * To derive clinical data to help inform the sample size for a future substantive study (the potential efficacy of additional on-line, patient education for SDD LH in achieving SDD compared to standard information giving).

Trial design and setting

Trial design:

A pilot, parallel, open, single centre, randomised controlled trial.

Trial Setting:

Recruitment to the Web-based Versus Standard Information for Same Day Hysterectomy (WISH) study will take place in gynaecology departments (general and relevant specialist clinics including menstrual disorders and pelvic pain clinics, hysteroscopy and colposcopy services) in an NHS, University-affiliated Teaching Hospital (Birmingham Women's & Children's Hospital (BWCH) in the UK.

Identification of participants:

Eligible women will be identified by a member of the clinical team responsible for the direct care of the potential participant in outpatient gynaecology clinics and pre-operative assessment clinics in each recruiting centre. Additionally, patients already on the waiting list for SDD LH will be identified and invited to participate. The study will be introduced by a member of the clinical or research team, with full counselling about the trial. The potential participant will be advised that participation in the study is entirely voluntary with the option of withdrawing from the study at any stage. It will be made clear that participation or non-participation will not affect their usual care.

Assessment of Risk:

SDD LH is routinely practiced at the BWCH. Verbal and written, paper-based information is provided. This study provides additional, on-line, multi-media information on a specifically designed website for SDD LH. Thus, this trial is categorised as: Type A = No higher than the risk of standard medical care.

Eligibility

Women are eligible for recruitment if they meet the inclusion criteria and do not have any of the exclusion criteria set out below:

Inclusion Criteria:

* Able to give informed consent to participate
* Have a benign gynaecological condition that is being treated with a LH
* Eligible to be on same day discharge pathway Patient factors

  * American Society of Anesthesiologists (ASA) physical status classification I/II with no sleep apnoea. ASA III may be suitable if comorbidities are stable and optimised.
  * No known cardio-pulmonary compromise
  * No known renal disease
  * Age </=60 years
  * BMI </=40
  * Not indication for admission to Gynaecological Extended Recovery Area (GERU) Surgical factors
  * Presumed benign disease
  * No anticipated surgical complications
  * Concomitant procedures acceptable but surgeon to decide on a case by case basis Discharge factors
  * Residence < 1 hour from BWCH
  * Access to transport from hospital to home

Exclusion Criteria:

* Patient above the age of 60
* Unwillingness or inability to comply with protocol procedures
* Women who require concomitant gynaecological surgery for bladder or other pelvic support
* Women who require concomitant gynaecological surgery for excision of deep endometriosis that requires dissection of the pararectal space

Consent

It will be the responsibility of the Investigator to obtain informed consent for each participant prior to performing any trial related procedure. A research nurse, research midwife or clinician is able to take consent providing that local practice allows this and responsibility has been delegated by the Principal Investigator as captured on the Site Signature and Delegation Log.

A Participant Information Sheet (PIS) will be provided to facilitate this process either at the time of initial consultation / hospital visit or sent through the post, via email, or by text as an attachment. Investigators or their delegate(s) will ensure that they adequately explain the aim, trial treatment, anticipated benefits and potential hazards of taking part in the trial to the participant. They will also stress that participation is voluntary and that the participant is free to decline to take part and may withdraw from the trial at any time. The participant will be given sufficient time to read the PIS and to discuss their participation with others outside of the site research team. The participant will be given the opportunity to ask questions. Where direct access to patient medical records is required the participant will give explicit consent for the regulatory authorities, members of the research team and or representatives of the sponsor to be given direct access to their medical records.

The Investigator or their delegate will then countersign and date the informed consent form (ICF). A copy of the ICF will be given to the participant (hard copy), a copy will be filed in the medical notes, and the original placed in the Investigator Site File (ISF). Once the participant is entered into the trial, the participant's trial number will be entered on the ICF maintained in the ISF.

Details of the informed consent discussions will be recorded in the participant's medical notes. This will include date of discussion, the name of the trial, summary of discussion, version number of the PIS given to participant and version number of ICF signed and date consent received. Where consent is obtained on the same day that the trial related assessments are due to start, a note should be made in the medical notes as to what time the consent was obtained and what time the procedures started.

Throughout the trial the participant will have the opportunity to ask questions about the trial. Any new information that may be relevant to the participant's continued participation will be provided. Where new information becomes available which may affect the participants' decision to continue, participants will be given time to consider and if happy to continue will be re-consented. Re-consent will be documented in the medical notes. The participant's right to withdraw from the trial at any time will remain.

Details of all patients approached about the trial will be recorded on the Participant Screening/Enrolment Log.

Recruitment, enrolment and randomisation

Recruitment:

Potential participants will be identified and approached by medical staff who are responsible for the direct care of the potential participant after having received appropriate training relating to the trial and who are delegated this task on the site delegation log. Recruitment will take place in gynaecology clinics in gynaecologist lead centres located across the United Kingdom.

The participant eligibility pathway to recruitment and randomisation is illustrated by the trial schema. Eligibility will be confirmed following discussions with the woman and a review of her medical notes by staff delegated this duty by the local principle investigator (PI).

Potential participants will be advised that taking part in the study is entirely voluntary and they may withdraw from the study at any stage without this affecting their usual care. Potential participants will be provided with a research ethics committee (REC) approved Study Participant Information Sheet (PIS) and given time to consider their involvement. However, as the intervention is simply an additional information resource (web-site link), patients will be allowed to consent during the initial consultation in clinic if they are willing to do so (PPI focus group felt that such an approach is acceptable because most women are comfortable with the internet and postal / phone follow up). However, as postal / phone follow up is required for up to 12 weeks, they will be made aware of this and take as much time as they need to consider participation.

Women who give consent will proceed to randomisation if they are eligible to participate in the trial. Consent will be recorded on the approved consent form, the original of which must be retained in the site file with a copy given to the participant.

Enrolment and Screening:

Women with benign gynaecological conditions requiring a LH and who are suitable for a SDD are eligible for inclusion. Prior to clinical consultations, the medical records of potential participants may be screened for eligibility by clinic doctors, nurses, research nurses and research midwives, after having received appropriate training relating to the trial. Clinic doctors will confirm eligibility for the trial. The same process will be applied to patients on the waiting list for SDD LH to identify eligible patients, contact them and invite them to participate.

Randomisation:

After participant eligibility has been confirmed and informed consent has been received, the participant can be randomised into the trial. Patients will be randomised in a 1:1 manner to either provision of the on-line SDD LH website resource (intervention) or standard practice for information provision (control). Randomisation will be performed via a web-based platform. If allocated to the intervention, then the website link will be provided in writing, via post, email or text (according to the patient's preference) immediately. Investigators will keep their own study file log which links patients with their allocated trial number in the trial Patient Recruitment and Identification Log.

Blinding:

Patients, clinicians, investigators, research assistants and responsible clinicians will not be blinded to the assigned allocation

Trial treatment / Intervention

Patients with a benign condition listed for a SDD LH agreeing to participate in the study who are allocated the intervention will be provided with the link to the SDD LH patient information website (see Table 1 and the website https://www.mydaycasehysterectomy.com). The option of this educational material will be in addition to the standard verbal and written patient information provided by the BWCH. Patients allocated the control group will receive standard BWCH information only.

The decision to remove or retain cervix (total or sub-total) or remove and retain ovaries will be left to the discretion of the participant in consultation with her gynaecologist. The LH will be performed or supervised by a surgeon who has self-declared as having expertise in laparoscopic hysterectomy and this requires the surgeon to meet minimum standards, regarding experience and case-load. Satisfactory experience will require surgeons to have performed a minimum of 30 cases and to have a current caseload of at least 12 cases per year

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent to participate
* Have a benign gynaecological condition that is being treated with a LH
* Eligible to be on same day discharge pathway Patient factors

  1. ASA I/II with no sleep apnoea. ASA III may be suitable if comorbidities are stable and optimised.
  2. No known cardio-pulmonary compromise
  3. No known renal disease
  4. Age </= 60 years
  5. BMI </=40
  6. Not indication for admission to Gynaecological Extended Recovery Area (GERU)
* Surgical factors

  1. Presumed benign disease
  2. No anticipated surgical complications
  3. Concomitant procedures acceptable but surgeon to decide on a case by case basis Discharge factors
  4. Residence < 1 hour from BWCH
  5. Access to transport from hospital to home

Exclusion Criteria:

* Patient above the age of 60
* Unwillingness or inability to comply with protocol procedures
* Women who require concomitant gynaecological surgery for bladder or other pelvic support
* Women who require concomitant gynaecological surgery for excision of deep endometriosis that requires dissection of the pararectal space above the age of 60
* Unwillingness or inability to comply with protocol procedures
* Women who require concomitant gynaecological surgery for bladder or other pelvic support
* Women who require concomitant gynaecological surgery for excision of deep endometriosis that requires dissection of the pararectal space

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Same Day Discharge following laparoscopic hysterectomy (0-23hours) | 0-24hours following surgery
  This means that the patient is discharged (leaves the hospital) before midnight on the day of surgery (case notes / electronic patient record).

SECONDARY OUTCOMES:
Satisfaction with care on discharge (bespoke patient questionnaire score) | 0-24hours following surgery
  Patient satisfaction of same day discharge following laparoscopic hysterectomy (LH). protocol. This will be assessed through bespoke patient questionnaire.
Acceptability and utility of patient education / information provided (score) | 6 weeks
  Patient satisfaction of acceptability and utility of patient education / information provided. This will be assessed through bespoke patient questionnaire.
Satisfaction with clinical outcome after laparoscopic hysterectomy (LH) (score) | 6 weeks
  Patient's satisfaction with clinical outcome after laparoscopic hysterectomy (LH) through(5-point Likert)
Satisfaction with care on discharge (score) | 6 weeks
  Patient's satisfaction with care on discharge through bespoke patient questionnaire
Generic quality of life post-surgery (score) | 6 weeks
  Patient's Quality of life score using EuroQol-5D-5L questionnaire
Generic quality of life post-surgery (score) | 6 weeks
  Patient's Quality of life score using EuroQol-5D-5L visual analogue scale
Contact with Community & Clinical Care Services | 6 weeks
  Serious Adverse Events through case report forms (CRF)
Time from surgery to resumption of usual activities in days | 6-12 weeks
  Time from surgery to resumption of usual activities using the PROMIS-SF (Patient-Reported Outcomes Measurement Information System Physical Function) questionnaire (item bank v1.2 will be used). Of the 29 items covering relevant activities for our study population, we have selected 8 items and. The selected items and the response categories were chosen by the PPI focus group to reflect the most common and generally applicable day-to-day activities. Participants will record when each activity is resumed, with full recovery being achieved once all 8 personalised activities have been resumed.
Time to return to work (if working) in days | 6-12 weeks
  This will be assessed using bespoke patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: TJustin Clark, MD, FRCOG, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared as part of results in a peer reviewed publication. No specific or individual participant data will be shared

REFERENCES:
- [Background] Lonky NM, Mohan Y, Chiu VY, Park J, Kivnick S, Hong C, Hudson SM. Hysterectomy for benign conditions: Complications relative to surgical approach and other variables that lead to post-operative readmission within 90 days of surgery. Womens Health (Lond). 2017 Aug;13(2):17-26. doi: 10.1177/1745505717714657. Epub 2017 Jun 29. PMID 28660800
- [Background] Madhvani K, Curnow T, Carpenter T. Route of hysterectomy: a retrospective, cohort study in English NHS Hospitals from 2011 to 2017. BJOG. 2019 May;126(6):795-802. doi: 10.1111/1471-0528.15539. Epub 2018 Dec 30. PMID 30461181
- [Background] Moawad G, Liu E, Song C, Fu AZ. Movement to outpatient hysterectomy for benign indications in the United States, 2008-2014. PLoS One. 2017 Nov 30;12(11):e0188812. doi: 10.1371/journal.pone.0188812. eCollection 2017. PMID 29190666
- [Background] Warren L, Ladapo JA, Borah BJ, Gunnarsson CL. Open abdominal versus laparoscopic and vaginal hysterectomy: analysis of a large United States payer measuring quality and cost of care. J Minim Invasive Gynecol. 2009 Sep-Oct;16(5):581-8. doi: 10.1016/j.jmig.2009.06.018. PMID 19835801
- [Background] Bailey CR, Ahuja M, Bartholomew K, Bew S, Forbes L, Lipp A, Montgomery J, Russon K, Potparic O, Stocker M. Guidelines for day-case surgery 2019: Guidelines from the Association of Anaesthetists and the British Association of Day Surgery. Anaesthesia. 2019 Jun;74(6):778-792. doi: 10.1111/anae.14639. Epub 2019 Apr 8. PMID 30963557
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, MacFie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):783-800. doi: 10.1016/j.clnu.2012.08.013. Epub 2012 Sep 28. PMID 23099039
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Perino A, Cucinella G, Venezia R, Castelli A, Cittadini E. Total laparoscopic hysterectomy versus total abdominal hysterectomy: an assessment of the learning curve in a prospective randomized study. Hum Reprod. 1999 Dec;14(12):2996-9. doi: 10.1093/humrep/14.12.2996. PMID 10601085
- See also: Related Info — https://www.mydaycasehysterectomy.com/
- See also: Related Info — https://www.gettingitrightfirsttime.co.uk/wp-content/uploads/2020/10/National-Day-Surgery-Delivery-Pack_Sept2020_final.pdf